CLINICAL TRIAL: NCT04402645
Title: Early Identification of Preterm Neonates With Evolving Chronic Pulmonary Hypertension: Utility of Functional Echocardiographic Markers
Brief Title: Novel Echocardiographic Methods for Early Identification of Neonates at Risk for Chronic Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Liverpool Women's NHS Foundation Trust (Other); The Rotunda Hospital (Other); University of Iowa (Other); BC Women's Hospital & Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 16-0111-E
Record Dates: First submitted 2020-05-13; First posted 2020-05-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Hypertension; Infant, Premature
Keywords: Premature Infant; Pulmonary Hypertension; Echocardiography; Extremely Low Birth Weight Neonate; Pulmonary Vascular Resistance; Right Ventricular Function
MeSH Terms: conditions — Hypertension, Pulmonary; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic pulmonary hypertension: Diagnosis on echocardiography at 36 weeks CGA using standard criteria (flat interventricular septal motion or right ventricular dilatation)
- No chronic pulmonary hypertension: Confirmed on echocardiography at 36 weeks CGA

SUMMARY:
Chronic pulmonary hypertension (cPHT) is a serious cardiopulmonary disorder that causes low oxygen levels in the blood, difficulty in breathing and ultimately heart failure. Newborn babies born extremely premature frequently suffer from cPHT while receiving treatment in neonatal intensive care units and are more likely to die than those without cPHT. Echocardiography is the investigation of choice for the assessment of heart function in premature infants however however there is a significant lack of standardization, sensitivity, and reliability for echocardiography parameters and a lack of consensus regarding optimal detection timing. In adults and older children it is known that early diagnosis and treatment, particularly before right side of the heart fails, is an important determinant of treatment success and survival. Diagnosis late in postnatal course for preterm infants remains a major barrier to timely and effective treatment.

The primary objective of this study is to develop new, sensitive, quantitative echocardiographic diagnostic criteria which will allow for the identification of extreme preterm neonates suffering from significantly high pressure in their pulmonary blood vessels, early in postnatal course, when the disease is likely to be most amenable to preventative/curative treatment.

This is an international initiative that will leverage expertise about echocardiography techniques and cardiopulmonary physiology of preterm infants.The results of this study will have an immediate impact on the day-to-day care of these highly vulnerable infants. The results will lead to increased awareness among clinicians, inform future surveillance protocols and diagnostic timing, and provide ideal preparation for future therapeutic trials.

DETAILED DESCRIPTION:
This is a multi-centre prospective observational study to develop new quantitative echocardiography diagnostic criteria sensitive to identify the presence of chronic pulmonary hypertension early in postnatal course. The investigators hypothesize that echocardiographic markers of pulmonary vascular resistance (PVR) and right ventricular (RV) function will allow early identification of extremely low birth weight (ELBW) preterm neonates who subsequently develop chronic pulmonary hypertension in association with chronic neonatal lung disease. More specifically, based on previous work and preliminary data, the investigators hypothesize that tricuspid annular plane systolic excursion (TAPSE- a routinely used marker of right heart function) and pulmonary artery acceleration time (PAAT- a routinely used marker of resistance in the pulmonary blood vessels) either alone or in combination will be the most sensitive parameters for early identification reducing the time to diagnosis compared to contemporary clinical practice.

The aim of the study is to recruit a large cohort of extreme premature neonates at two weeks of age and sequentially perform two "early-diagnostic assessments". First assessment will be performed between 14-21 days of life and the second at a corrected gestational age (CGA) of 32 weeks. Assessment will include a focused ultrasound of the heart to measure pre-defined markers which are under investigation. The investigators will test the diagnostic utility of these markers separately for each time point. All babies will also have a standard diagnostic assessment for evaluation of cPHT at 36 weeks CGA, as per routine practice. The study team will record this data for participants, along with their relevant medical details and clinical outcomes, including neurodevelopment assessments performed at 18 months of age as a routine clinical follow-up. At the end of this study, the investigators will divide the cohort into those who developed cPHT and those who did not as per currently used standard criteria and will compare the results of new parameters obtained at earlier time points. The sensitivity of each marker to pick-up early cPHT will be calculated and its correlation with health outcomes will be established.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth ≤26+6/7 and/or birth weight <1000g
* Alive at two weeks of postnatal age
* Infant cleared by the clinical team for approach

Exclusion Criteria:

* Known major congenital and/or genetic anomaly
* Congenital heart defects (CHD) except patent ductus arteriosus (PDA), patent foramen ovale (PFO), peripheral pulmonary artery stenosis and small (< 3 mm in diameter) ventricular septal defects
* Any condition which, in the opinion of the investigator, would preclude enrollment

Min Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants will be recruited from tertiary neonatal intensive care units (NICUs) in Toronto (Mount Sinai Hospital and Sunnybrook Health Sciences Centre) and Vancouver (BC Women's Hospital & Health Centre) Canada, the United States (University of Iowa Health Care, Iowa), and Europe (Liverpool University Hospitals NHS Foundation Trust and The Rotunda Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic test characteristics calculated for TAPSE and PAAT against diagnosis of chronic pulmonary hypertension on standard diagnostic assessment | Early diagnostic assessments (14-21 days postnatal age; 32+0/7-32+6/7); Standard diagnostic assessment (~36 weeks CGA)
  Sensitivity, specificity, positive and negative likelihood ratios for TAPSE and PAAT at each early diagnostic assessment against diagnosis of chronic pulmonary hypertension on standard diagnostic assessment using echocardiography using current standard criteria

SECONDARY OUTCOMES:
Composite of Death/ Chronic Neonatal Lung Disease | Composite outcome measure will be assessed on the date of discharge for each study participant from the study Neonatal Intensive Care Unit (NICU) or date of death during admission (if applicable) up to 365 days.
  Infant death prior to 36 weeks CGA and chronic neonatal lung disease are competing risks for the primary outcome of chronic pulmonary hypertension. The presence of both will be assessed.
Duration of need for respiratory support | Outcome measure will be assessed on the date of discharge for each study participant from the study Neonatal Intensive Care Unit (NICU) or date of death during admission (if applicable) up to 365 days.
  Total duration of need (number of days) for invasive, non-invasive and supplemental (low-flow) oxygen support
Length of hospital stay | Outcome measure will be assessed on the date of discharge for each study participant from the study Neonatal Intensive Care Unit (NICU) or date of death during admission (if applicable) up to 365 days.
  Length of NICU admission from birth to discharge (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Amish Jain, MD, PHD, Principal Investigator — Staff Neonatologist, Clinician Scientist
Locations (6):
- University of Iowa Health Care, Iowa City, Iowa, United States
- Canada (3):
  - BC Women's Hospital & Health Centre, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
- Rotunda Hospital, Dublin, Ireland
- Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas L, Baczynski M, Deshpande P, Kharrat A, Joye S, Zhu F, Ibarra-Rios D, Shah PS, Mertens L, Jankov RP, Ye XY, Neary E, Ting J, Castaldo M, Levy P, Smith A, El-Khuffash AF, Giesinger RE, McNamara PJ, Weisz DE, Jain A. Multicentre prospective observational study exploring the predictive value of functional echocardiographic indices for early identification of preterm neonates at risk of developing chronic pulmonary hypertension secondary to chronic neonatal lung disease. BMJ Open. 2021 Mar 31;11(3):e044924. doi: 10.1136/bmjopen-2020-044924. PMID 33789855